#### The GlaxoSmithKline group of companies

209635

| Division | : | Worldwide Development |
|------------------|---|---------------------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) Amendment |

Title : Reporting and Analysis Plan for a randomized, double-blind, single ascending dose study to determine the safety and tolerability, pharmacokinetics and pharmacodynamics of GSK3772847 administered subcutaneously in healthy participants

Compound Number : GSK3772847

Clinical Study : 209635

Identifier : Refer to Document Date

#### **Description:**

The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 209635 (Document Number 2020N427367\_02).

This RAP is intended to describe the safety, tolerability, pharmacokinetics and pharmacodynamics analyses required for the study.

This RAP will be provided to the study team members to convey the content of Statistical Analysis Complete (SAC) deliverables.

This version of the RAP includes amendments to the originally approved RAP.

## **RAP Author(s):**

| Author |
|---|
| Lead |
| PPD |
| Principal Statistician (Respiratory, Clinical Statistics) |
| <b>Co-Authors</b> |
| PPD |
| Programming Leader (Clinical Programming, Respiratory) |
| PPD |
| Pharmacokinetics (Respiratory, Clinical Pharmacology Modelling and Simulation) |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

209635

#### **RAP Team Reviews:**

# RAP Team Review Confirmations (Method: E-mail)



# Clinical Statistics & Clinical Programming Line Approvals (Method: e-signature)

| Approver |
|--------------------------------------------------------|
| PPD , |
| Statistics Director (Respiratory, Clinical Statistics |
| PPD |
| Programming Manger (Respiratory, Clinical Programming) |

209635

# **TABLE OF CONTENTS**

| | | PAGE |
|---|---|---|
| 1. | INTRODUCTION | 6 |
| | 1.1. RAP Amendments | 6 |
| 2. | SUMMARY OF KEY PROTOCOL INFORMATION | 6 |
| | 2.1. Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. Study Objective(s) and Endpoint(s) | |
| | 2.3. Study Design | 9 |
| | 2.4. Statistical Hypotheses | 10 |
| 3. | PLANNED ANALYSES | 11 |
| | 3.1. Instream Review and Interim Analyses | |
| | 3.2. Final Analyses | |
| 4. | ANALYSIS POPULATIONS | 12 |
| | 4.1. Protocol Deviations | 13 |
| 5. | CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONVENTIONS | 14 |
| | 5.1. Study Treatment & Sub-group Display Descriptors | 14 |
| | 5.2. Baseline Definitions | 15 |
| | 5.3. Examination of Covariates, Other Strata and Subgroups | 16 |
| | 5.3.1. Strata | 16 |
| | 5.4. Other Considerations for Data Analyses and Data Handling Conventions | 16 |
| 6. | STUDY POPULATION ANALYSES | 17 |
| <b>7</b> . | EFFICACY ANALYSES | 18 |
| 8. | SAFETY ANALYSES | 19 |
| | 8.1. Adverse Events Analyses | |
| | 8.2. Adverse Events of Special Interest Analyses | |
| | 8.3. Clinical Laboratory Analyses | |
| | 8.4. COVID-19 Displays | 19 |
| 9. | PHARMACOKINETIC ANALYSES | 21 |
| | 9.1. Primary Pharmacokinetic Analyses | 21 |
| | 9.1.1. Endpoint / Variables | 21 |
| | 9.1.1.1. Drug Concentration Measures | |
| | 9.1.1.2. Derived Pharmacokinetic Parameters | 21 |
| | 9.1.2. Summary Measure | |
| | 9.1.3. Population of Interest | |
| | 9.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | 9.1.5. Statistical Analyses / Methods | 22 |
| 10. | POPULATION PHARMACOKINETIC (POPPK) ANALYSES | 23 |
| 11. | PHARMACODYNAMIC ANALYSES | 23 |
| | 11.1 Secondary Pharmacodynamic Analyses | |

209635

Endpoint / Variables 23 11.1.1. 11.1.2. Summary Measure ......23 Population of Interest 23 11.1.3. 11.1.4. 11.1.5. 12.1.1. 12.1.2. Population of Interest 24 12.1.3. Strategy for Intercurrent (Post-Randomization) Events ......24 12.1.4. 12.1.5. 14 REFERENCES 26 15.2. 15.3. Appendix 4: Study Phases and Treatment Emergent Adverse 15.4. 15.4.2. 15.5. 15.5.1. 15.5.2. 15.5.3. 15.6. 15.6.1. General 37 15.6.2. Safety 37 15.6.3. 15.6.4. 15.7. 15.7.1. 15.7.2. 15.8. Appendix 9: Population Pharmacokinetic (PopPK) Analyses ................42 15.11. Appendix 11: List of Data Displays.......45 15.11.1. Data Display Numbering .......45 

 15.11.4. Study Population Tables
 46

 15.11.5. Safety Tables
 48

 15.11.6. Pharmacokinetic Tables
 52

 15.11.7. Pharmacodynamic Tables
 53

 15.11.8. Pharmacokinetic: Figures
 55

 15.11.9. Pharmacodynamic Figures
 57

 15.11.10. ICH Listings
 60

 15.11.11. Non-ICH Listings
 63

 15.12. Appendix 12: Example Mock Shells for Data Displays
 65

209635

## 1. INTRODUCTION

| The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol Revision Chronology | | |
|---|---|---|
| 2020N427367_02 | | |
| 2020N427367_01 | 12/JUN/2020 | Amendment 1 |
| 2020N427367_00 17/MAR/2020 Original | | |

Amendment 1 includes a COVID-19 measures appendix, increased outpatient visit windows and defines a sample collection window for free sST2 and total sST2 blood samples.

Amendment 2 reduces the age range from 18-65 to 18-50 to ensure older populations, potentially more at risk of COVID-19 are not recruited into the study and to update secondary pharmacodynamics endpoint to specify nominal day as maximum timepoint.

#### 1.1. RAP Amendments

- To drop interim analysis due to the termination of aIL33r clinical development
- To remove some of the data displays due to the termination of aIL33r clinical development
- To add Covid-19 related data displays
- To remove 'Randomised Population' from Section 4. Analysis Population because this population is not used in any data display.

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| The PKPD population | The PKPD population has been defined as two separate populations (A PK and PD population) | Having two separate populations will make things clearer. For example if a subject has a PK sample taken, but no PD sample and vice versa. |
| Section 9.4.3 Maximal decrease from baseline in free sST2 and maximal increase from baseline in total | The formal analysis has been removed but the endpoint will still be summarised. | Comparisons with placebo are not of interest |

209635

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| soluble sST2 levels in serum will be analysed. | | The impact of injection site is of key interest (which will not be assessed in an ANCOVA analysis given the small numbers per cohort per injection site). The results for percent suppression from the summary tables will be reported in the CSR (and not from an analysis). |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | Primary |
| To evaluate the safety and tolerability of a single dose of GSK3772847, compared with placebo administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants. | Occurrence of adverse events (AEs) and serious adverse events (SAEs) (including injection site reactions) |
| To assess the pharmacokinetics (PK) of a single dose of GSK3772847 administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants (Cohorts 1 and 2 also summarised by injection site) | PK parameters, including but not limited to, Area under<br>the plasma-concentration time curve (AUC), maximum<br>plasma concentration (Cmax), time to Cmax (Tmax) and<br>terminal half-life (t1/2) of GSK3772847 per cohort.<br>(Cohorts 1 and 2 also summarised by injection site) |
| Secondary | Secondary |
| To evaluate the pharmacodynamics (PD) of a single dose of GSK3772847 administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants. | <ul> <li>Maximal decrease from baseline in free soluble ST2 levels in serum up to a maximum of 85 days post dose</li> <li>Maximal increase from baseline in total soluble ST2 levels in serum up to a maximum of 85 days post dose</li> </ul> |
| To assess the immunogenicity of a<br>single dose of GSK3772847<br>administered subcutaneously in<br>healthy participants including cohorts<br>of Japanese and Chinese participants. | Occurrence of anti-GSK3772847 antibodies |
| To assess potential changes in<br>Cytochrome P450 3A4 (CYP3A4)<br>enzyme activity following a single<br>dose of GSK3772847in healthy<br>participants including cohorts of<br>Japanese and Chinese participants. | Plasma 4β-Hydroxycholesterol (4βOH) /cholesterol ratio as an endogenous marker for CYP3A4 activity pretreatment and following a single dose of GSK3772847 |

| Objectives | Endpoints |
|---|---|
| Other | Other |
| To further assess the safety and tolerability of a single dose of GSK3772847, compared with placebo administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants. | <ul> <li>12-lead electrocardiogram (ECG) measurements</li> <li>Clinical chemistry laboratory tests</li> <li>Vital signs</li> </ul> |
| To evaluate the pharmacodynamics (PD) of a single dose of GSK3772847 administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants. | <ul> <li>Free and total soluble ST2 levels in serum</li> <li>Blood eosinophil levels</li> </ul> |
| To assess the pharmacokinetics (PK) of a single dose of GSK3772847 administered subcutaneously in healthy participants including cohorts of Japanese and Chinese participants | GSK3772847 levels in serum |

209635

# 2.3. Study Design



209635

| Overview of Study Design and Key Features | | | | |
|---|---|---|---|---|
| | 1,2 | G | Placebo SC | Abdomen |
| | 1,2 | Н | Placebo SC | Thigh |
| | 1,2,3 | I | Placebo SC | Upper Arm |
| | and 4 | | | |

# 2.4. Statistical Hypotheses

The primary objective of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK3772847 administered subcutaneously. There are no formal hypothesis tests associated with this objective and no formal significance tests. The information acquired from this study will be used to quantify the effects of GSK3772847 on safety and tolerability via the SC route where the main focus will be on injection site reactions and to assess the pharmacokinetics and pharmacodynamics across the 3 injection sites and doses. In addition, PK will be evaluated in Japanese and Chinese participants.

209635

## 3. PLANNED ANALYSES

# 3.1. Instream Review and Interim Analyses

A dose escalation committee will review blinded summary safety data (including injection site data obtained up to 48 hours post-dose) of at least 20 participants from cohort 1.

The Dose Escalation charter will describe the procedures related to DEC operations in greater detail. The dose escalation committee (DEC), comprised of members from the GSK Study Team (namely safety and clinical) and the Investigator(s), will review blinded safety data (including injection site data obtained 48 hours post-dose) from at least 20 participants in cohort 1 before initiating dosing in cohorts 2, 3 and 4. Dose escalation may occur only after review of individual injection site data. The decision to proceed to dosing in cohorts 2, 3 and 4 will be made by the Dose Escalation Committee based on assessment of the injection site data at 70mg dose level. Data may be reviewed in an unblinded fashion by a subset of the DEC (namely safety and clinical) should a significant safety concern arise during the blinded review.

An interim analysis was originally planned to inform on the properties of GSK3772847 dosed via the subcutaneous route and allow the project to move forward to the next phase of development. Due to the termination of aIL33r clinical development, this interim analysis is no longer needed.

# 3.2. Final Analyses

The final planned primary analyses will be performed according to IQVIA's procedures after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in Section 4.4 of the protocol: A participant is considered to have completed the study if he/she has completed all phases of the study including the final follow up visit.
- 2. All required database cleaning activities have been completed and final soft lock), and final database lock) have been declared by Data Management. IQVIA final database lock is defined as no changes can be made to the data and the end of the study milestone has been reached with all data clean, SDV'd, frozen and locked.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to IQVIA procedures using SAS v9.4.
- 5. Final SDTM sent to GSK (defined as GSK final DBF)

209635

# 4. ANALYSIS POPULATIONS

The following populations (as defined below), will include participants who are randomized and replaced because they withdraw prior to D29:

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | All participants who sign the ICF | Study Population |
| Pharmacokinetic | The PK population consists of all randomized subjects who received at least one dose of study treatment, and for whom at least one post-randomisation pharmacokinetic sample was obtained, analyzed and was measurable. Displays will be based on the treatment and injection site which the participant actually received. | PK outputs |
| Pharmacodynamic | The PD population consists of all randomized subjects who received at least one dose of study treatment, and for whom at least one pharmacodynamic sample was obtained, analyzed and was measurable. Displays will be based on the treatment and injection site which the participant actually received. | PD outputs |
| Safety | All randomized participants who take at least 1 dose of study intervention. Participants will be analyzed according to the treatment they actually received. | Study Population Safety |

Refer to 15.11 Appendix 11: List of Data Displays which details the population used for each display.

209635

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, participant management or participant assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team and IQVIA throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This output will be based on data as recorded on the inclusion/exclusion page of the eCRF.

209635

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | | | |
|---|---|---|---|---|---|
| Treat | ment Description in | randomisation | Data Displays for Reporting | | |
| Code | Description | Injection Site | Description | Injection Site | Order in TLF |
| А | 70mg SC<br>GSK3772847 /<br>Abdomen | Abdomen | 70mg SC<br>GSK3772847 | Abdomen | 2 |
| В | 70mg SC<br>GSK3772847/<br>Thigh | Thigh | 70mg SC<br>GSK3772847 | Thigh | 3 |
| С | 70mg SC<br>GSK3772847 /<br>Upper Arm | Upper Arm | 70mg SC<br>GSK3772847 | Upper Arm | 4 |
| D | 140mg SC<br>GSK3772847 /<br>Abdomen | Abdomen | 140mg SC<br>GSK3772847 | Abdomen | 6 |
| E | 140mg SC<br>GSK3772847 /<br>Thigh | Thigh | 140mg SC<br>GSK3772847 | Thigh | 7 |
| F | 140mg SC<br>GSK3772847 /<br>Upper Arm | Upper Arm | 140mg SC<br>GSK3772847 | Upper Arm | 8 |
| G <sup>2</sup> | Placebo SC /<br>Abdomen | Abdomen | Placebo SC | Abdomen | NA |
| H <sup>2</sup> | Placebo SC /<br>Thigh | Thigh | Placebo SC | Thigh | NA |
| <b> </b> 2 | Placebo SC /<br>Upper Arm | Upper Arm | Placebo SC | Upper Arm | NA |
| J <sup>1</sup> | 70mg SC<br>GSK3772847 | Overall (Cohort 1) | 70mg SC<br>GSK3772847<br>Overall | Combined (Cohort 1) | 5 |
| K¹ | 140mg SC<br>GSK3772847 | Overall (Cohort 2) | 140mg SC<br>GSK3772847<br>Overall | Combined (Cohort 2) | 9 |
| L | 140mg SC<br>GSK3772847/<br>Upper Arm | Upper Arm | Japanese<br>140mg SC<br>GSK3772847 | Upper Arm | 11 |
| М | 140mg SC<br>GSK3772847/<br>Upper Arm | Upper Arm | Chinese140m<br>g SC<br>GSK3772847 | Upper Arm | 12 |
| N¹ | Placebo SC | Overall (Cohorts 1 and 2) | Placebo SC | Combined(Co<br>horts 1 &2) | 1 |

209635

| | Treatment Group Descriptions | | | | |
|---|---|---|---|---|---|
| Treat | ment Description in | randomisation | Dat | a Displays for R | leporting |
| Code | Description | Injection Site | Description | Injection Site | Order in TLF |
| O <sup>1</sup> | Placebo SC | Overall (Cohorts 3 and 4) | Placebo SC | Combined(Co<br>horts 3&4) | 10 |

<sup>1</sup>J, K, N and O will not be received in the randomisation file, and will be derived within the AdAM datasets.

For summary tables, Cohorts 1 and 2 will be summarised overall (i.e. by treatment and across all injection sites), in addition to per injection site. Placebo data will be pooled across injection site for cohorts 1 and 2 and similarly across Japanese and Chinese participants for cohorts 3 and 4.

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Assessments | Considered a | s Baseline | Baseline Used in |
|---|---|---|---|---|
| | Screening | Day 0 | Day 1 (Pre-<br>Dose) | Data Display |
| Safety | | | | |
| Vital Signs | X | X | Х | Day 1 (Pre-Dose) |
| 12-lead Electrocardiogram (ECG) measurements | Х | | X | Day 1 (Pre-Dose) |
| Clinical laboratory<br>tests (haematology<br>and chemistry) | X | | Х | Day 1 (Pre-Dose) |
| Pharmacokinetic | | | | |
| PK Blood samples | | | Χ | Day 1 (Pre-Dose) |
| Pharmacodynamic | | | | |
| Free sST2 and total sST2 blood sample | | | X | Day 1 (Pre-Dose) |
| Biomarker | | | | |
| Immunogenicity:<br>Anti-GSK3772847<br>antibodies | | | X | Day 1 (Pre-Dose) |
| Plasma 4βOH cholesterol | | | Х | Day 1 (Pre-Dose) |

<sup>&</sup>lt;sup>2</sup>G, H are for cohorts 1 and 2 only and I is for cohorts 1,2, 3 and 4.

209635

Unless otherwise stated, if baseline data is missing, the latest assessment pre-dose will be used.

# 5.3. Examination of Covariates, Other Strata and Subgroups

## 5.3.1. Strata

The list of strata may be used in descriptive summaries. Additional strata of clinical interest may also be considered.

| Category | Details |
|----------|--------------------------------------------|
| Stratum | Injection site for all summary statistics. |

# 5.4. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 15.3 | Appendix 3: Assessment Windows |
| 15.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 15.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 15.6 | Appendix 6: Derived and Transformed Data |
| 15.7 | Appendix 7: Reporting Standards for Missing Data |
| 15.8 | Appendix 8: Values of Potential Clinical Importance |

209635

# 6. STUDY POPULATION ANALYSES

The study population analyses will be based on the Safety population, unless otherwise specified. Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

209635

# 7. EFFICACY ANALYSES

There are no efficacy analyses to be included in this study.

209635

## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified.

## 8.1. Adverse Events Analyses

The definition of an AE is detailed in Appendix 3 of the protocol.

Separate analyses of AEs will be conducted including those events that are captured during the on-treatment period as well as the post-treatment period defined in Section 15.4.

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting. The updated GSK respiratory Adverse Events of Special Interest (AESIs) can be found in the following folder (aesi.sas7bdat):

\\uk1salx00175.corpnet2.com\arenv\arprod\respiratory\res\_safety\aesi\refdata.

The details of the planned displays are provided in Appendix 11: List of Data Displays.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests (including blood eosinophil levels), Urinalysis, and Liver function tests will be based on GSK Core Data Standards. Clinical laboratory summaries will include all assessments post-baseline. The laboratory assessments for each category are displayed below (Table 4 in Section 10.2 of Appendix 2 of the protocol):

## 8.4. COVID-19 Displays

Due to the short duration and small size of the study, only listings will be produced for COVID-19 related data. The details of the planned COVID-19 displays are in Appendix 11: List of Data Displays.

209635

Table 2 Protocol-Required Safety Laboratory Assessments

| Laboratory<br>Assessments | Parameters | | | | |
|---|---|---|---|---|---|
| Haematology | Platelet Count | t | RBC<br>Indices: | | count with Differential otnote 3): |
| | RBC Count | | MCV | WBC | |
| | | | | Neutro | phils |
| | Haemoglobin | | MCHC | Lymph | ocytes |
| | Haematocrit | | | Monoc | |
| | | | | Eosino | |
| | | | | Basoph | nils |
| Clinical<br>Chemistry | BUN | Potassium | AST (SGOT) | | Total and direct bilirubin |
| | Creatinine | Sodium | ALT (SGPT) | | Total Protein |
| | Glucose | Calcium | Alkaline phosphatase | | Albumin |
| | | Magnesium | | | |
| Routine<br>Urinalysis | Microscop | se, protein, b<br>pic examinat | | R (if blo | lipstick od or protein is haematuria of $\geq 1+]$ ) |
| Other tests | • hsCRP | | | | |
| Other | • HIV | | | | |
| Screening | • Hepatitis | В | | | |
| Tests | - | C (Hep C an | • / | | |
| | • FSH and estradiol (as appropriate) | | | | |
| | <ul> <li>Alcohol, cotinine and drug screen (to include at minimum:<br/>amphetamines, barbiturates, cocaine, opiates, cannabinoids and<br/>benzodiazepines)</li> </ul> | | | | |

Abbreviations: ALT (SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT) = aspartate aminotransferase (serum glutamic oxaloacetic transaminase); BUN = blood urea nitrogen; FSH = follicle stimulating hormone; HBsAg = hepatitis B surface antigen; anti-HBc = hepatitis B core antibody; hsCRP = highly sensitive C-reactive protein; MCHC = mean corpuscular haemoglobin concentration; MCV = mean corpuscular volume; RBC = red blood cell; UACR = urinary albumin-creatinine ratio; WBC = white blood cell, pH= hydrogen ion concentration.

- 1. Details of liver chemistry stopping criteria and required actions and follow-up assessments after liver stopping or monitoring event are given in Section 7.1 and Appendix 6 (of the protocol). All events of ALT ≥3 × upper limit of normal (ULN) and bilirubin ≥2 × ULN (>35% direct bilirubin) or ALT ≥3 × ULN and international normalized ratio (INR) >1.5, if INR measured, which may indicate severe liver injury (possible Hy's Law), must be reported as an SAE (excluding studies of hepatic impairment or cirrhosis).
- 2. Local urine testing will be standard for the protocol unless serum testing is required by local regulation or IRB/IEC.
- 3. WBC differentials will be reviewed at screening only, in order to confirm participant eligibility. At all other times the site must order haematology test with blinded differentials.

209635

## 9. PHARMACOKINETIC ANALYSES

# 9.1. Primary Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 15.5.3 Reporting Standards for Pharmacokinetic)

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic (PK)" population, unless otherwise specified.

Plasma concentrations will be listed and summarised by cohort. Cohorts 1 and 2 will also be summarised by injection site. See Section 9.1.2 for details on the summary measures used.

Refer to the PK Guidance document, titled Non-Compartmental Analysis of Pharmacokinetic Data (GUI\_51487) for more information regarding the treatment of concentrations below the assay's lower limit of quantification (NQ).

The details of the planned displays are presented in Appendix 11: List of Data Displays

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the plasma-concentration time curve from time zero to the time of last quantifiable concentration (C(t)). |
| | Calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the plasma-concentration time curve from time zero extrapolated to infinite time. |
| Cmax | Maximum observed concentration. |
| | Determined directly from the concentration-time data. |
| tmax | Time to Cmax of GSK3772847 |
| t1/2 | Terminal half-life of GSK3772847 will be calculated as |
| | • t1/2 = ln2 / lambda_z |
| %AUCext | The percentage of AUC(0-∞) obtained by extrapolation (%AUCex) will be calculated |
| | as: |
| | • [AUC(0-∞) – AUC(0-t)] / AUC(0-∞) x 100 |

209635

| Parameter | Parameter Description |
|---|---|
| Ct | The last observed quantifiable concentration |
| Tlast | Time of last quantifiable concentration |
| * associated pa | * associated parameters lambda_z, lambda_z_lower, lambda_x_upper, No_points_lambda_z to be listed. NOTES: |
| Additional parameters may be included as required. Lambda_z is the terminal phase rate constant. | |

## 9.1.2. Summary Measure

Descriptive statistics will be calculated by cohort for all PK concentrations over time and for the derived PK parameters. Additionally, for cohorts 1 and 2 parameters will be summarised per injection site.

• For each of the PK derived parameters AUC (0-inf), AUC (0-t), t1/2 and Cmax, the following summary statistics will be calculated and tabulated: N, n, Geometric Mean, %CV, Min, Median, Max.

For tmax, the summary statistics shall include N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum.

• For PK concentration data, the following summary statistics will be calculated and tabulated by treatment: N, n, arithmetic mean, 95% confidence interval (CI), SD, median, minimum, Q1. Q3, maximum

### 9.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the PK population, unless otherwise specified.

#### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

No intercurrent events are defined for this study. All data collected for each participant in the relevant population will be included in the analysis.

• Missing and anomalous concentration data not due to intercurrent events will be handled by CPMS according to SOP\_314000.

## 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

209635

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Population PKPD analyses may be conducted using data from this study as part of a multi-study analyses to inform on the PK and PD properties of GSK3772847 and will not have any impact on the conduct or reporting of study 209635. These analyses will be conducted by CPMS, if conducted, and will be reported separately so will not be described in this RAP.

# 11. PHARMACODYNAMIC ANALYSES

# 11.1. Secondary Pharmacodynamic Analyses

## 11.1.1. Endpoint / Variables

- Maximal decrease from baseline in free soluble ST2 levels in serum
- Maximal increase from baseline in total soluble ST2 levels in serum

## 11.1.2. Summary Measure

Change from baseline in free and total soluble ST2 levels in serum will be calculated in the ADaM (Analysis Data Model) Datasets (see Section 15.6.4 for derivation)

Maximal decrease from baseline in free sST2 and maximal increase from baseline in total soluble sST2 levels in serum will be summarised and listed.

Descriptive statistics will be calculated by cohort for maximal decrease from baseline in free sST2 and maximal increase in total soluble sST2. Additionally, for cohorts 1 and 2 parameters will be summarised per injection site.

For maximal decrease from baseline in free sST2 and maximal increase in total soluble sST2 data, the following summary statistics will be calculated and tabulated: n, Geometric Mean, %CV, Min., Q1. Q3, Median, Max

#### 11.1.3. Population of Interest

The secondary pharmacodynamics analyses will be based on the PD population, unless otherwise specified.

#### 11.1.4. Strategy for Intercurrent (Post-Randomization) Events

No intercurrent events are defined for this study. All data collected for each participant in the relevant population will be included in the analysis.

209635

### 11.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 11.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 12. BIOMARKER ANALYSES

## 12.1. Biomarker Analyses

### 12.1.1. Endpoint / Variables

Incidence and prevalence of anti-GSK3772847 antibodies and Plasma 4βOH /cholesterol ratio (pre-treatment and following dosing of GSK3772847).

# 12.1.2. Summary Measure

Summaries of the incidence of and titres of anti- GSK3772847 antibodies on Day 1 (predose), 15, 29, 57, 85 will be produced.

The plasma  $4\beta$ OH/cholesterol ratio will be calculated at each visit in the ADaM datasets. Change from baseline will be summarised as a ratio to the pre-treatment visit i.e using the following derivation: post-dosing of GSK3772847/ pre-treatment). Samples post-dose will be received on Days 5, 15, 29 and 85. Pre-treatment sample will be taken Day 1 pre-dose.

#### 12.1.3. Population of Interest

The biomarker analyses will be based on the PD population, unless otherwise specified.

#### 12.1.4. Strategy for Intercurrent (Post-Randomization) Events

No intercurrent events are defined for this study. All data collected for each participant in the relevant population will be included in the analysis.

# 12.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 11.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

209635

## 13. OTHER ENDPOINTS

12-Lead ECGs, clinical laboratory safety tests, vital signs, blood eosinophil levels, free and total soluble sST2 levels in serum and GSK3772847 levels in the serum will be listed and summarised by cohort (and injection site for cohorts 1 and 2) over time.

# 13.1. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 11: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, blood eosinophil levels and free and total soluble sST2 levels in serum and GSK3772847 levels in the serum will be summarised using descriptive statistics (n, Geometric Mean, %CV, Min., Q1. Q3, Median, Max (95% CIs will be included for ratio to baseline) and Geometric mean and 95% CI graphically presented (where appropriate) and listed.

12-Lead ECGs, and vital signs will be summarised using descriptive statistics (n, Arithmetic Mean, SD, Median, Min and Max) and listed.

209635

# 14. REFERENCES

GlaxoSmithKline Document Number 2020N427367\_02, Protocol: A randomized, double-blind, single ascending dose study to determine the safety and tolerability, pharmacokinetics and pharmacodynamics of GSK3772847 administered subcutaneously in healthy participants [02/JUL/2020].

Protocol Deviation Management Plan (PDMP) [09/JUN/2020]

209635

## 15. APPENDICES

# 15.1. Appendix 1: Exclusions from Per Protocol Population

Instream and final analysis population reviews as per SOP 130050 are not planned for this study because it does not include a Per-Protocol population.

However, protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan. Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset. This dataset will be the basis for the summaries and listings of protocol deviations.

209635

# 15.2. Appendix 2: Schedule of Activities

# 15.2.1. Protocol Defined Schedule of Events

| | | Da | y 1 ( | Hour | s) | | | | | | | | | | | | | | Notes<br>Time window for |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>0 | Pre-<br>dose | 0 | 2 | 4 | 8 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>9 | Day<br>15 | Day<br>29 | Day<br>43 | Day<br>57 | Day<br>71 | Day<br>85/Early<br>withdrawal<br>visit | Outpatient visits: Day $9\pm2$ , Day $15\pm4$ days, and Days 29, 43 and $57\pm7$ days, Days 71 and $85\pm10$ days |
| Clinic Visits | | | | | | | | | | | | | | | | | | | |
| Admission to clinic | Х | | | | | | | | | | | | | | | | | | Participants may remain in the clinic until day 6 with visits at days 6-8 as outpatient, at the investigator's discretion |
| Inclusion/Exclusion criteria review | Х | | | | | | | | | | | | | | | | | | |
| Discharge from clinic | | | | | | | | | | | Х | | | | | | | | |
| Out-patient visit | | | | | | | | | | | | Χ | Χ | Χ | Χ | Χ | Χ | Х | |
| Study Intervention | | | | | | | | | | | | | | | | | | | |
| Randomisation | | Χ | | | | | | | | | | | | | | | | | |
| SC dosing | | | Х | | | | | | | | | | | | | | | | |
| Safety<br>Assessments | | | | | | | | | | | | | | | | | | | |
| Safety labs<br>(haematology,<br>clinical chemistry<br>and urinalysis) | | X | | | | | Х | | Х | | | Х | | Х | Х | | | X | WBC differentials<br>MUST be blinded<br>(see Appendix 2 in<br>protocol) |

| | | Da | y 1 ( | Hour | rs) | | | | | | | | | | | | | | Notes<br>Time window for |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>0 | Pre-<br>dose | 0 | 2 | 4 | 8 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>9 | Day<br>15 | Day<br>29 | Day<br>43 | Day<br>57 | Day<br>71 | Day<br>85/Early<br>withdrawal<br>visit | Outpatient visits:<br>Day $9 \pm 2$ , Day $15 \pm 4$ days, and Days $29$ ,<br>$43$ and $57 \pm 7$ days,<br>Days 71 and $85 \pm 10$<br>days |
| | | | | | | | | | | | | | | | | | | | To be taken in non-<br>fasted state |
| Alcohol/drug screen | Χ | | | | | | | | | | | | | | | | | | |
| Urinary Cotinine<br>Test | Х | | | | | | | | | | | | | | | | | | |
| 12-lead ECG | | Х | | | | Х | | Х | | Х | | | | Х | | Х | | Х | When scheduled at<br>the same timepoint,<br>ECG's should be<br>taken as close as<br>possible to PK<br>samples |
| Vital signs | Х | Х | | | | Х | Х | Х | Х | Х | Х | | | Х | | Х | | х | Supine blood<br>pressure and heart<br>rate |
| Concomitant medications | <b>▼</b> === | ====== | === | | ==== | ==== | ===== | ===== | ===== | ===== | ==== | ===== | ===== | ==== | ===== | ===== | ==== | ====== | |
| SAE/AE Review | <b>▼</b> | | ==== | -=== | ==== | ==== | ===== | ===== | ===== | ===== | ===== | | ===== | ===== | ===== | ===== | ===== | ====== | Including injection site reactions |

| | | Da | y 1 (l | Hour | s) | | | | | | | | | | | | | | Notes<br>Time window for |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>0 | Pre-<br>dose | 0 | 2 | 4 | 8 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>9 | Day<br>15 | Day<br>29 | Day<br>43 | Day<br>57 | Day<br>71 | Day<br>85/Early<br>withdrawal<br>visit | Outpatient visits:<br>Day $9 \pm 2$ , Day $15 \pm 4$ days, and Days 29,<br>43 and $57 \pm 7$ days,<br>Days 71 and $85 \pm 10$<br>days |
| Local Injection site reaction evaluation | | | | | X | | X | X | | | | | | | | | | | Targeted evaluation at 4 hours post-dose on Day 1 & 24 hours post-dose on Day 2 and 48 hours post-dose on Day 3. Spontaneous reporting at all other times. |
| Pregnancy test | Х | | | | | | | | | | | | | Χ | | X | | X | Serum pregnancy test<br>at screening and urine<br>dipstick test at all<br>other visits |
| Brief Physical<br>Examination | | | | | | | | | | | | | | | | | | X | |
| Biomarker<br>Collection | | | | | | | | _ | | | | | | | | | | | |
| PK blood sample | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Day 1 samples +/- 1<br>hours. Days 2-6 +/- 2<br>hours relative to time<br>of dosing |

| | | Da | y 1 (l | Hour | s) | | | | | | | | | | | | | | Notes<br>Time window for |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Day<br>0 | Pre-<br>dose | 0 | 2 | 4 | 8 | Day<br>2 | Day<br>3 | Day<br>4 | Day<br>5 | Day<br>6 | Day<br>9 | Day<br>15 | Day<br>29 | Day<br>43 | Day<br>57 | Day<br>71 | Day<br>85/Early<br>withdrawal<br>visit | Outpatient visits:<br>Day $9 \pm 2$ , Day $15 \pm 4$ days, and Days 29,<br>43 and $57 \pm 7$ days,<br>Days 71 and $85 \pm 10$<br>days |
| Free sSt2 and total sST2 blood sample | | Х | | Х | Х | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Χ | Х | Samples should be taken within ± 2 |
| Immunogenicity blood sample | | Х | | | | | | | | | | | Х | Х | | Х | | Х | minutes of PK Collect pre-dose on Day 1 |
| 4βOH<br>cholesterol/choleste<br>rol plasma sample | | Х | | | | | | | | Х | | | Х | Х | | | | Х | All samples should be in non-fasted state for comparison with baseline. |
| Pharmacogenetic (PGx) blood sample | | | | Х | | | | | | | | | | | | | | | May be taken at any time post-dose |

- The timing and number of planned study assessments, including safety, pharmacokinetic, pharmacodynamic/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments as the result of emerging pharmacokinetic/pharmacodynamic data from this study must be documented and approved by the relevant study team member and then archived in the sponsor and site study files but will not constitute a protocol amendment. The Competent Authority (CA) and ethics committee (EC) will be informed of any safety issues that constitute a substantial amendment and require alteration of the safety monitoring scheme or amendment of the informed consent form (ICF). The changes will be approved by the CA and the EC before implementation.
- When scheduled at the same timepoints, vital signs should be conducted followed by ECG's prior to any blood draws.

209635

# 15.3. Appendix 3: Assessment Windows

### 15.3.1. Definitions of Assessment Windows for Analyses

Dosing should occur up to 28 days after screening.

No assessment windows will be defined for Day 0, Day 1 (pre-dose), Day 1 2hrs, Day 1 4hrs, Day 1 8hrs, Day 2, Day 3, Day 4, Day 5 and Day 6 analyses. Summaries and analyses will be based on nominal visits as these are inpatient visits.

For the following outpatient visits, assessment windows are as follows:

- Day  $9 \pm 2$  days
- Days  $15 \pm 4$  days
- Days 29, 43,  $57 \pm 7$  days
- Days, 71 and  $85 \pm 10$  days.

If two visit dates overlap then the assessment that is closest to the scheduled visit is assigned as that visit assessment and the other visit would be assigned as an unscheduled visit e.g. if a subject has a day 9 visit outside the day 9 window but is in the window of the day 15 visit then the visit closest to day 15 gets assigned to day 15 and the other visit becomes an unscheduled visit.

Analysis will be performed on actual time (for adverse events) and nominal time for all other endpoints. No exclusion will be made to plasma samples taken outside the sample windows as long as there is time recorded. Any data falling outside of these assessment windows will be classified as unscheduled visits

209635

# 15.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

# 15.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to dose.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Start Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date + 28 days |
| Post-Treatment | Date > Study Treatment Stop Date + 28 days |

# 15.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
| Pre-treatment | <ul> <li>Conmed Start Date &lt; Study Treatment First Dose Date</li> <li>Conmed End Date &lt; Study Treatment First Dose Date</li> <li>CMSTRF = "BEFORE"</li> <li>Randomisation date is missing i.e. subject was not randomised</li> </ul> |
| On-treatment | <ul> <li>Study Treatment First Dose Date &lt;= Conmed Start Date &lt;= Study Treatment Last Dose Date + 28</li> <li>Study Treatment First Dose Date &lt;= Conmed End Date &lt;= Study Treatment Last Dose Date + 28</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(Conmed Start Date &lt;= Study Treatment Last Dose Date + 28) and (CMENRF ="DURING/AFTER" or CMENRF ="AFTER" or CMSTRF = "DURING")</li> <li>(CMSTRF = "BEFORE" or CMSTRF = "DURING" or CMENRF = "DURING/AFTER") and (Conmed End Date &gt;= Study Treatment First Dose Date)</li> <li>(CMSTRF = "BEFORE" or CMSTRF ="DURING") and (CMENRF = "DURING/AFTER" or CMENRF = "AFTER")</li> <li>CMSTRF = "DURING"</li> <li>CMSTRF = "DURING/AFTER"</li> </ul> |
| Post-treatment | <ul> <li>Conmed Start Date &gt; Study Treatment Last Dose Date + 28</li> <li>Conmed End Date &gt; Study Treatment Last Dose Date + 28</li> <li>CMENRF = "AFTER"</li> <li>CMENRF = "DURING/AFTER"</li> </ul> |
| All phases | Conmed start date is missing and CMSTRF is missing and conmed end date is missing and CMENRF is missing |

209635

| Study Phase | Definition Note: All programming should use start and end dates where available, CMSTRF and CMENRF are only to be used where dates are unavailable to help determine the correct study phase. |
|---|---|
|---|---|

#### 1. NOTES:

- The duration of a single concomitant medication can extend over multiple study phases
- Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

# 15.4.2. Treatment Emergent Flag for Adverse Events

Adverse Events will be flagged as Treatment Emergent as described in the table in Section 15.4.1, where the AE Start Date/Time will be considered. If the study treatment stop date is missing, then the AE will be considered to be on-treatment.

209635

# 15.5. Appendix 5: Data Display Standards & Handling Conventions

# 15.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : UK1SALX00175 |
| HARP Compound | : the following directories will be used for the final analysis: |
| | : \arprod\gsk3772847\mid209635\final_01 |
| Analysis Datasets | |
| Analysis datasets will be created according to CDISC standards (SDTM Implementation Guide Version 3.2 & AdaM Implementation Guide Version 1.1. | |
| Generation of RTF Files | |
| <ul> <li>RTF files will be generated for all tables in the final reporting effort for use in writing the<br/>CSR.</li> </ul> | |

# 15.5.2. Reporting Standards

#### General

- The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
  - Do not include participant level listings in the main body of the GSK Clinical Study Report. All
    participant level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

209635

| Unscheduled Visits | |
|---|---|
| Unscheduled visits will only be included in summary tables as part of 'minimum/maximum post baseline' and 'minimum/maximum change from baseline' summary. | |
| Unscheduled visits will not be included in figures. | |
| All unscheduled visits will be included in listings. | |
| Descriptive Summary Statistics | |
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to GSK Standard Statistical Display Principals 7.01 to 7.13. | |

# 15.5.3. Reporting Standards for Pharmacokinetic

| Reporting of Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive | Refer to IDSL PK Display Standards. |
| Summary Statistics | Refer to IDSL Statistical Principle 6.06.1. |
| , | Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Reporting of Pharm | Reporting of Pharmacokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, and between geometric coefficient of variation (CVb (%)), Min, Median, Max will be reported. $ CV_b \ (\%) = \sqrt{\left( exp(SD^2) - 1 \right) * 100} $ (SD = SD of log transformed data) |
| Parameters Not<br>Being Log<br>Transformed | $T_{max},T_{last},$ first point, last point, and number of points used in the determination of $\lambda z,\% AUCex$ |
| Summary Tables | All provided PK parameters will be summarised except Lamz, lamzUL, LamzLL, LamzNP and AUC % extrapolated area , Rsq-adjusted (if calculated). |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |
209635

#### 15.6. Appendix 6: Derived and Transformed Data

#### 15.6.1. General

#### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 15.3.1) the value closest to the target
  day for that window will be used. If values are the same distance from the target, then the mean will
  be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

#### 15.6.2. Study Population

#### Age

- Only year of birth will be collected on the CRF and birth date will be presented in listings as 'YYYY'.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as '30th June' and then calculated based on the dose date.

#### 15.6.3. Safety

#### **ECG Parameters**

#### **Laboratory Parameters**

If a laboratory value which is expected to have a numeric value for summary purposes, has a nondetectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

- Example 1: 2 Significant Digits  $\rightarrow$  '< x'becomes x -0.01
- Example 2: 1 Significant Digit  $\rightarrow$ '> x' becomes x + 0.1
- Example 3: 0 Significant Digits  $\rightarrow$  '< x' becomes x -1

209635

#### 15.6.4. Pharmacodynamic and Biomarker

#### Free and Soluble ST2

#### Maximal decrease in free/Maximal Increase in total Soluble ST2 from baseline

Change from baseline in free soluble ST2 levels in serum will be calculated in the ADaM (Analysis Data Model) Datasets as follows for each individual for all assessments:

Free soluble ST2 in serum assessment at Timepoint X – Baseline

For all timepoints (X) post dose where a free soluble ST2 in serum assessment has been taken and Baseline is defined in Section 5.2. Maximal decrease from baseline is then the largest decrease calculated across all timepoints post dose. Maximum increase from baseline in total soluble ST2 level will be calculated in a similar manner albeit as the largest increase from baseline.

#### Plasma 4βOH /cholesterol ratio

The plasma  $4\beta$ OH/cholesterol ratio will be calculated for each visit in the ADaM datasets. Change from baseline will be summarised as a ratio to the pre-treatment visit i.e. using the following derivation: post-dosing of GSK3772847/ pre-treatment). Samples post-dose will be received on Days 5, 15, 29 and 85. Pre-treatment sample will be taken Day 1 pre-dose.

See also Section 12.1.1

209635

### 15.7. Appendix 7: Reporting Standards for Missing Data

### 15.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | For the final analysis, participant study completion (i.e. as specified in the protocol) is defined as having completed all phases of the study including the final follow up visit. Participants who will be explaned in the actual Participants. |
| | Participants who withdraw prior to D29 will be replaced in the study. Replacement participants will be dosed with the planned treatment of the withdrawn participant. |
| | All available data from participants including those who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| | The Withdrawal visit will be slotted as per Appendix 3: Assessment Windows or will be summarised as the withdrawal visit. |

### 15.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| | <ul> <li>No manual imputation will be made for any missing numerical data.</li> </ul> |
| | <ul> <li>Missing data will generally not be considered in the calculation of percentages<br/>(i.e., the denominator will not include subjects who have missing data at a given<br/>time point).</li> </ul> |
| Outliers | Any participants excluded from the summaries will be documented along with the reason for exclusion in the clinical study report. |

### 15.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: |
| | Missing Start Day: First of the month will be used unless this is before the start<br>date of study treatment; in this case the study treatment start date will be used and<br>hence the event is considered On-treatment as per Appendix 4: Study Phases and<br>Treatment Emergent Adverse Events. |
| | <ul> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop<br/>date of study treatment; in this case the study treatment stop date will be used.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | The recorded partial date will be displayed in listings. |

209635

### 15.8. Appendix 8: Values of Potential Clinical Importance

Values of potential clinical importance will not be used in this study, instead normal reference ranges of "Low", "Normal" and "High" will be used.

209635

### 15.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

Population PKPD analyses may be conducted using data from this study as part of a multi-study analyses to inform on the PK and PD properties of GSK3772847 and will not have any impact on study 209635. These analyses will be conducted by CPMS and will be reported separately so will not be described in this RAP.

209635

## 15.10. Appendix 10: Abbreviations & Trademarks

## 15.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| AUC(0-∞) | Area under the plasma concentration-time curve, from time zero to infinity |
| AUC(0-t) | Area under the plasma concentration-time curve, from time zero to the time of |
| , | the last quantifiable concentration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library (GSK Standards Library) |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |

209635

| Abbreviation | Description |
|--------------|--------------------------------------------|
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SDV | Source Data Verification |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| Tmax | Time to Cmax |
| t1/2 | Apparent terminal phase half-life |

## 15.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| IQVIA |
| NONMEM |
| SAS |
| WinNonlin |

209635

#### 15.11. Appendix 11: List of Data Displays

All displays (Tables, Figures & Listings) will use the term 'Subjects' instead of "Participants".

#### 15.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-----------------------|------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Safety | 2.1 to 2.n 2.1 to 2.n | |
| Pharmacokinetic | 3.1 to 3.n 3.1 to 3.n | |
| Pharmacodynamic | 4.1 to 4.n | 4.1 to 4.n |
| Biomarker | 5.1 to 5.n | 5.1 to 5.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

#### 15.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic or Biomarker | PD_Fn | PD_Tn | PD_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 15.11.3. Deliverables

| Delivery [Priority] | Description |
|---------------------|-------------------------------------|
| Final SAC | Final Statistical Analysis Complete |

209635

# 15.11.4. Study Population Tables

| Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| Subject | Disposition | | | | | |
| 1.1. | Safety | ES8 | Summary of Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | Final<br>SAC | Prog |
| 1.2. | ASE | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements Note that the reasons for rescreen of subjects who initially failed but subsequently entered the study are not included in the display. This will be footnoted. | Final<br>SAC | Prog |
| Populat | ion Analysed | | | | | |
| 1.3. | ASE | SP1 | Summary of Study Populations | IDSL | Final<br>SAC | Prog |
| Demog | raphic and Bas | eline Characteris | tics | | | |
| 1.4. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | Final<br>SAC | Prog |
| 1.5. | ASE | DM11 | Summary of Age Ranges | EudraCT | Final<br>SAC | Prog |
| 1.6. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | Final<br>SAC | Prog |

| Study Population Tables | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| Prior ar | nd Concomitan | t Medications | | | | |
| 1.7. | Safety | MH4 | Summary of Current Medical Conditions at Screening | ICH E3 | Final<br>SAC | Prog |
| 1.8. | Safety | SU1 | Summary of Smoking History at Screening | | Final<br>SAC | Prog |

209635

# 15.11.5. Safety Tables

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| Advers | e Events (AEs) | | | | | |
| 2.1. | Safety | SAFE_T01 | Overview of On-treatment Adverse Events During the Study | See 3.01 /arenv/arprod/gsk3772847/mid207597/fi nal_02/output for example Include footnote defining "On- treatment" | Final<br>SAC | Prog |
| 2.2 | Safety | SAFE_T01 | Overview of Post-treatment Adverse Events During the Study | Include footnote defining "Post-treatment" | Final<br>SAC | Prog |
| 2.3 | Safety | AE1 | Summary of All On-treatment Adverse Events by System Organ Class and Preferred Term | ICH E3. Include footnote defining "Ontreatment" See 3.02 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.4 | Safety | AE1 | Summary of All Post-treatment Adverse Events by System<br>Organ Class and Preferred Term | ICH E3. Include footnote defining "Post-treatment" See 3.02 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.5 | Safety | AE1 | Summary of All On-treatment Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | ICH E3. Include footnote defining "Ontreatment" | Final<br>SAC | Prog |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| 2.6 | Safety | AE1 | Summary of All On-treatment Fatal Adverse Events by System Organ Class and Preferred Term | ICH E3. Include footnote defining "Ontreatment" See 3.07 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.7 | Safety | AE3 | Summary of All On-treatment Common (>=1%) Adverse Events by Overall Frequency | ICH E3. Include footnote defining "Ontreatment" See 3.08 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.8 | Safety | AE1 | Summary of On-treatment Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 See 3.09 /arenv/arprod/gsk3772847/mid207597/fi nal_02/output for example. Include footnote defining "Ontreatment" | Final<br>SAC | Prog |
| 2.9 | Safety | AE15 | Summary of All On-treatment Common (>=1%) Non-serious<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | FDAAA, EudraCT. Include footnote defining "On-treatment" See 3.10 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| 2.10 | Safety | AE1 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | Include footnote defining "On-<br>treatment" See 3.11 /arenv/arprod/gsk3772847/mid207597/fi<br>nal_02/output for example | Final<br>SAC | Prog |
| 2.11 | Safety | AE16 | Summary of All On-treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of<br>Participants and Occurrences) | FDAAA, EudraCT. Include footnote defining "Ontreatment" See 3.13 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.13 | Safety | AE1 | Summary of All On-treatment Serious Adverse Events Leading to Withdrawal from Study by System Organ Class and Preferred Term | IDSL. Include footnote defining "Ontreatment" See 3.15 /arenv/arprod/gsk3772847/mid207597/final_02/output for example | Final<br>SAC | Prog |
| 2.14 | Safety | AE1 | Summary of On-treatment Injection Site Reactions | A subset of 3.03 where we display the injection site reactions only. Include footnote defining "On-treatment" | Final<br>SAC | Prog |
| Advers | e Events of Spe | ecial Interest (AES | Sis) | | | |
| 2.15 | Safety | AE1 | Summary of On-treatment Adverse Events of Special Interest | IDSL | Final<br>SAC | Prog |
| 2.16 | Safety | LB1 | Summary of Clinical Chemistry | ICH E3 | Final<br>SAC | Prog |

| Safety: | Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Delive<br>rable<br>[Priori<br>ty] | Stats<br>or<br>Prog |
| 2.17 | Safety | LB1 | Summary of Change from Baseline in Clinical Chemistry | ICH E3 | Final<br>SAC | Prog |
| 2.18 | Safety | LB1 | Summary of Hematology | ICH E3 | Final<br>SAC | Prog |
| 2.19 | Safety | LB1 | Summary of Changes from Baseline in Hematology | ICH E3 | Final<br>SAC | Prog |
| 2.20 | Safety | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | Final<br>SAC | Prog |
| 2.21 | Safety | EG1 | Summary of ECG Findings | IDSL | Final<br>SAC | Prog |
| 2.22 | Safety | VS1 | Summary of Vital Signs | ICH E3 | Final<br>SAC | Prog |
| 2.23 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | Final<br>SAC | Prog |

209635

## 15.11.6. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| Second | Secondary: Pharmacokinetic | | | | | |
| 3.1 | PK | PK01 | Summary of GSK3772847 Serum Concentration-Time Data (ug/ml) by Cohort, and Injection Site | The display will be summarised by the following: | Final SAC | Prog |
| 3.2 | PK | PK04 | Summary of Derived GSK3772847 Pharmacokinetic Parameters by Cohort, and Injection Site | | Final SAC | Prog |

209635

# 15.11.7. Pharmacodynamic Tables

| Phar | macodynamic | c Tables | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| Seco | ndary Pharm | acodynamic: Free an | d Total SST2 | | | |
| 4.1 | PD | Table 6.01 CSR:<br>2019N414678_00<br>207597 | Summary of Raw and Change from Baseline in Free Soluble ST2 concentration (ng/mL) by Cohort and Injection Site | The display will be summarised by the following treatment groups: 70 mg dose abdomen injection site 70 mg dose thigh injection site 70 mg dose arm injection site Cohort 1 140 mg dose abdomen injection site 140 mg dose thigh injection site 140 mg dose arm injection Cohort 2 Cohort 3 140 mg Japanese population Cohort 4 140 mg Chinese population Placebo (pooled Cohorts 1+2) Placebo (pooled Cohorts 3+4) Include a line for maximum increase from baseline (for all treatments) | Final SAC | Prog |
| 4.2 | PD | Table 6.09 CSR:<br>2019N414678_00<br>207597 | Summary of Raw and Change from Baseline in Total Soluble ST2 concentration (ng/mL) by Cohort and Injection Site | The display will be summarised by the following treatment groups below • 70 mg dose abdomen injection site • 70 mg dose thigh injection site • 70 mg dose arm injection site • Cohort 1 • 140 mg dose abdomen injection site • 140 mg dose thigh injection site | Final SAC | Prog |

| Phar | rmacodynamic | Tables | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| | | | | <ul> <li>140 mg dose arm injection</li> <li>Cohort 2</li> <li>Cohort 3 140 mg Japanese population</li> <li>Cohort 4 140 mg Chinese population</li> <li>Placebo (pooled Cohorts 1+2)</li> <li>Placebo (pooled Cohorts 3+4)</li> <li>Include a line for maximum decrease from baseline (for all treatments)</li> </ul> | | |
| 4.3 | PD | | Summary of Observed Results and Change from baseline in Plasma 4β hydroxycholesterol /cholesterol ratio | See t_4_06(002).pdf in med_ds_proj/\Projects\Respiratory & Inflammation\GSK3772847 (IL33)\209635\RAP\TFLs | Final SAC | |
| 4.4 | PD | | Summary of Incidence and Titres of Anti-<br>GSK3772847 Antibodies | See Table 4.02<br>'arenv/arprod/gsk3772847/207597/final_02/output' | Final SAC | |

209635

# 15.11.8. Pharmacokinetic: Figures

| Pharm | Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| Secon | Secondary: Pharmacokinetic | | | | | |
| 3.1 | PK | | Serum Concentrations of GSK3772847 over Time by Dose and Injection Site | Plot median and range PK concentration over time. There will be 2 plots. One for cohort 1 (70mg) and one for cohort 2 (140mg). Each plot will have 3 groups of different line type differentiating between the injection sites Cohort dose abdomen injection site Cohort dose thigh injection site Cohort dose arm injection site | Final SAC | Prog |
| 3.2 | PK | | Serum Concentrations of GSK3772847 over Time by Ethnicity for 140 mg SC Dose | Plot median and range PK concentration over time. There will be 3 groups of different line type. Cohort 2 (upper arm injection site) Cohort 3 (Japanese population) Cohort 4 (Chinese population) Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |

| Pharm | Pharmacokinetic Figures | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| 3.3 | PK | | Serum Concentrations of GSK3772847 over Time by Dose | Plot median and range PK concentration over time. There will be 2 groups of different line type. One for cohort 1 (70mg) and one for cohort 2 (140mg). Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |

209635

# 15.11.9. Pharmacodynamic Figures

| Pharma | codynamic: Figure | s | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| Seconda | Secondary: Pharmacodynamic | | | | | |
| 4.1 | PD | | Free Soluble ST2 levels by Dose, Injection Site and Placebo | Plot median and range free sst2 over time. There will be 2 plots. One for cohort 1 (70mg) and one for cohort 2 (140mg). Each plot will have 4 groups of different line type differentiating between the injection sites Cohort dose abdomen injection site Cohort dose thigh injection site Cohort dose arm injection site Placebo (pooled Cohorts 1+2) Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |
| 4.2 | PD | | Free Soluble ST2 levels by Ethnicity and Placebo for 140 mg SC Dose | Plot median and range free sst2 over time. There will be 5 groups of different line type. Cohort 2 (upper arm injection site) Cohort 3 (Japanese population) Cohort 4 (Chinese population) Placebo (pooled Cohorts 1+2) Placebo (pooled Cohorts 3+4) Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |

| Pharma | codynamic: Figure | es | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| 4.3 | PD | | Free Soluble ST2 levels by Dose and Placebo | Plot median and range free sST2 over time. There will be 3 groups of different line type: cohort 1 (70mg) cohort 2 (140mg) placebo (pooled Cohorts 1+2). Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |
| 4.4 | PD | | Total Soluble ST2 levels by Dose, Injection Site and Placebo | Plot median and range total sst2 over time. There will be 2 plots. One for cohort 1 (70mg) and one for cohort 2 (140mg). Each plot will have 4 groups of different line type differentiating between the injection sites Cohort dose abdomen injection site Cohort dose thigh injection site Cohort dose arm injection site Placebo (pooled Cohorts 1+2) Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |

| Pharmacodynamic: Figures | | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | Stats<br>or<br>Prog |
| 4.5 | PD | | Total Soluble ST2 levels by Ethnicity and Placebo for 140 mg SC Dose | Plot median and range total sst2 over time. There will be 5 groups of different line type. Cohort 2 (upper arm injection site) Cohort 3 (Japanese population) Cohort 4 (Chinese population) Placebo (pooled Cohorts 1+2) Placebo (pooled Cohorts 3+4) Plot on normal and logarithmic (base10) scales. | Final SAC | Prog |
| 4.6 | PD | | Total Soluble ST2 levels by Dose and Placebo | Plot median and range total sST2 over time. There will be 3 groups of different line type: | Final SAC | Prog |

209635

# 15.11.10. ICH Listings

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen and Run-in Failure | Journal Guidelines | Final SAC |
| 2. | Safety | ES2 / ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | Final SAC |
| 3. | Safety | BL1 / BL2 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | Final SAC |
| 4. | Safety | TA1 /<br>CP_RD1x | Listing of Planned and Actual Treatments | IDSL | Final SAC |
| Protoc | Protocol Deviations | | | | |
| 5. | Safety | DV2 | Listing of Important Protocol Deviations | ICH E3 | Final SAC |
| 6. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | Final SAC |
| Demog | Demographic and Baseline Characteristics | | | | |
| 7. | Safety | DM2 | Listing of Demographic Characteristics | ICH E3 | Final SAC |
| 8. | Safety | DM9 | Listing of Race | ICH E3 | Final SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitar | nt Medications | | , | |
| 9. | Safety | CP_CM3 | Listing of Concomitant Medications | IDSL | Final SAC |
| Exposi | ure and Treatm | ent Compliance | | | |
| 10. | Safety | EX3 | Listing of Exposure Data | ICH E3 | Final SAC |
| Advers | se Events | | | | |
| 11. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | Final SAC |
| 12. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | Final SAC |
| 13. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study | ICH E3 | Final SAC |
| 14. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | Final SAC |
| Seriou | s and Other Sig | nificant Adverse | Events | | |
| 15. | Safety | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | Final SAC |
| 16. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | Final SAC |
| 17. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | Final SAC |
| 18. | Safety | AE8 | Listing of Serious Adverse Events Leading to Withdrawal from Study | ICH E3 | Final SAC |
| 19. | Safety | AE8 | Listing of Adverse Events of Special Interest | ICH E3 | Final SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Hepato | biliary (Liver) | | | | |
| 20. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | Final SAC |
| 21. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | Final SAC |
| All Lab | oratory | | | | |
| 22. | Safety | LB5 / LB6 | Listing of All Laboratory Data for Participants with Any Value Outside Normal Range | ICH E3 | Final SAC |
| 23. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | Final SAC |
| ECG | | | | | • |
| 24. | Safety | EG5 | Listing of All ECG Findings for Participants with an Abnormal ECG Finding | IDSL | Final SAC |
| 25. | Safety | EG5 | Listing of Abnormal ECG Findings | IDSL | Final SAC |
| Vital Si | gns | | | | |
| 26. | Safety | VS4 | Listing of All Vital Signs Data | IDSL | Final SAC |

209635

# 15.11.11. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 27. | Safety | ESI8 | Listing of AE Terms of Special Interest | IDSL | Final SAC |
| Liver E | vents: Note on | ly produced if the | re is a Liver Event | | |
| 28. | Safety | LIVER5 | Listing of Liver Events | | Final SAC |
| 29. | Safety | LIVER6 | Listing of Liver Event Information for RUCAM Score | | Final SAC |
| 30. | Safety | LIVER7 | Listing of Liver Biopsy | | Final SAC |
| 31. | Safety | LIVER8 | Listing of Liver Imaging Details | | Final SAC |
| Cardio | vascular Event | s: Note only prod | uced if there is a Cardiovascular Event | | |
| 32. | Safety | Patient Profile | Listing of Myocardial infarction/unstable angina | | Final SAC |
| 33. | Safety | Patient Profile | Listing of Congestive heart failure | | Final SAC |
| 34. | Safety | Patient Profile | Listing of Arrhythmias | | Final SAC |
| 35. | Safety | Patient Profile | Listing of Valvulopathy | | Final SAC |
| 36. | Safety | Patient Profile | Listing of Pulmonary hypertension | | Final SAC |
| 37. | Safety | Patient Profile | Listing of Cerebrovascular events/stroke and transient ischemic attack | | Final SAC |
| 38. | Safety | Patient Profile | Listing of Peripheral arterial thromboembolism | | Final SAC |
| 39. | Safety | Patient Profile | Listing of Deep venous thrombosis/pulmonary embolism | | Final SAC |
| 40. | Safety | Patient Profile | Listing of Revascularisation | | Final SAC |
| 41. | Safety | Patient Profile | Listing of Deaths | | Final SAC |

| Pharmo | ockinetics | | | |
|---|---|---|---|---|
| 42. | PK | | Listing of GSK3772847 Plasma Pharmacokinetic Concentration – Time Data | Final SAC |
| 43. | PK | | Listing of Derived GSK3772847 Plasma Pharmacokinetic Parameters | Final SAC |
| Pharma | acodynamics | | | , |
| 44. | PD | | Listing of Free and Total Soluble ST2 Concentrations | Final SAC |
| 45. | PD | | Listing of Maximum decrease from baseline in Free and Maximum increase from baseline in Total Soluble ST2 Concentrations | Final SAC |
| 46. | PD | | Listing of Plasma 4β hydroxycholesterol/cholesterol ratio | Final SAC |
| 47. | PD | | Listing of Anti-GSK3772847 Antibodies | Final SAC |
| 48. | PD | | Listing of Blood Eosinophil Data | Final SAC |
| Covid- | 19 | | | |
| 49. | Safety | PAN7 | Listing of All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic | Final SAC |
| 50. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom<br>Assessments for Subjects with COVID-19 Adverse Events | Final SAC |
| 51. | Safety | DV2 | Listing of Non-Important COVID-19 related Protocol Deviations | Final SAC |

209635

## 15.12. Appendix 12: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request

## Signature Page for 209635 TMF-6054409 v1.0

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: 04-Dec-2020 14:13:34 GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Author Date of signature: 09-Dec-2020 10:15:53 GMT+0000 |

Signature Page for TMF-6054409 v1.0